CLINICAL TRIAL: NCT06300528
Title: PERFORM: A Phase II Study of Pemigatinib in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphomas
Brief Title: Pemigatinib in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI181541
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: All Patients (Experimental): The study will investigate the effectiveness of pemigatinib.
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib will be self-administered as a once-a-day oral treatment on a 28-day cycle.
  Other Names: Pemazyre

SUMMARY:
The purpose of this clinical trial is to learn if the study drug pemigatinib is effective in treating patients with relapsed or refractory B-cell non-Hodgkin lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years.
* ECOG Performance Status ≤ 2.
* Histologically confirmed MCL or MZL, including EMZL/MALT lymphoma, SMZL, and NMZL.

  --Patients with gastric MALT lymphoma and those who are H. Pylori positive need to have failed a trial of H. Pylori eradication and are either ineligible, have refused, or have failed gastric radiation therapy.
* Have received at least two prior lines of systemic therapy and do not have FDA approved available therapies or have refused them.
* Prior autologous hematopoietic cell transplantation (auto-HCT) and CAR-T cell therapy are eligible.

  * Patients with prior auto-HCT may be eligible if treatment completed after at least 3 months prior to first treatment
  * Patients with CAR T-cell therapy may be eligible if treatment completed after at least 1 month prior to first treatment
* Subject must have an indication for systemic treatment.
* Radiographically measurable disease by computed tomography (CT) scan, defined as at least one lesion >1.5 cm in size or assessable disease in the opinion of the investigator.
* Life expectancy >3 months, in the opinion of the investigator.
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥ 1000/mm3 (≥1.0 x 10^9/L) independent of G-CSF support (i.e., no G-CSF within the past 3 days), unless there is documented bone marrow involvement or splenomegaly with ensuing cytopenia in which case ANC of 750 cells/mm3 (0.75 x 10^9/L) is permissible. Also, there should be no evidence of myelodysplasia or hypoplastic bone marrow.
    * Platelet count ≥ 75,000/mm3 (≥75 x 10^9/L) independent of transfusion support (i.e., no transfusion within the past 3 days) unless there is documented bone marrow involvement in which case platelet count of 50,000 cells/mm3 (0.5 x 10^9/L) is permissible. Patients must be responsive to transfusion support if given for thrombocytopenia and patients refractory to transfusion support are not eligible. Also, there should be no evidence of myelodysplasia or hypoplastic bone marrow.
    * Hemoglobin ≥ 8 g/dL independent of transfusion support (i.e., no transfusion within the past 3 days) unless there is documented bone marrow involvement or splenomegaly with ensuing cytopenia in which case hemoglobin of 7 g/dL is permissible. Patients must be responsive to transfusion support if given for anemia and patients refractory to transfusion support are not eligible. Also, there should be no evidence of myelodysplasia or hypoplastic bone marrow.
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN). or <2.5 x ULN with document liver involvement and/ or Gilbert's disease
    * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN ----Subjects with liver involvement will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.
    * Renal:

      ----Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula.
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    ---Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and

    ---Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or

    ---Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Female subjects of childbearing potential and male subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.3.1.
* Ability to swallow oral tablets.
* Recovery to baseline or ≤ Grade 2 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy per the treating investigator.
* Patients or their legal representatives must be able to read, understand, and provide informed consent to participate in the trial.

Exclusion Criteria:

* Prior receipt of FGFR inhibitor.
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of the study drug.
* Concurrent anticancer therapy except as listed in section 6.7.2 for prostate and breast cancer.
* Prior systemic anti-cancer therapy or any investigational therapy within the timeframes listed below:

  * Cytotoxic chemotherapy within 4 weeks prior to treatment.
  * Monoclonal antibody within 3 weeks prior to treatment
  * BTK inhibitor within 2 weeks prior to treatment. ---Note: The wash out interval is based on the last day of the prior therapy to the start of the study drug (C1D1).
* Prior radiotherapy within 4 weeks prior to the first dose of study treatment.

  --Note: Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have radiation pneumonitis. A 2-week washout is permitted for palliative radiation to non-CNS disease.
* Major surgery 4 weeks prior to starting study drug or who have not fully recovered from major surgery.
* Active second malignancy which is expected to impact study participation, in the opinion of the investigator.
* Known CNS involvement.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  --Cardiovascular disorders:
  * Congestive heart failure New York Heart Association Class III or IV or serious cardiac arrhythmias.
  * Unstable angina pectoris or acute coronary syndrome within the past 2 months prior to study enrolment
  * History of myocardial infarction (MI) within 3 months prior to enrollment.
  * QTcF prolongation defined as a QTcF > 470 ms

    * Correction of suspected drug induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation.
    * Correction for underlying bundle branch block (BBB) allowed.
    * Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker.
    * Left ventricular ejection fraction < 40% in the 12 months prior to study enrollment
    * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the drug through a feeding tube], etc.)
* Known HIV infection.
* Active hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.

  --Note: Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects with SMZL who have chronic HCV will need to have undergone antiviral treatment to participate.
* History and/or current evidence of ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, myocardia, or lung, excepting calcified lymph nodes and asymptomatic arterial or cartilage/tendon calcification.
* Current evidence of clinically significant corneal or retinal disorder confirmed by ophthalmologic examination
* Use of any potent CYP3A4 inhibitors or inducers or moderate CYP3A4 inducers within 14 days or 5 half-lives (whichever is longer) before the first dose of study drug. Moderate CYP3A4 inhibitors are not prohibited but should be avoided.
* Subject with history of hypovitaminosis D requiring supraphysiologic dose (such as 50,000 IU of vitamin D3) to replenish the deficiency. Subjects receiving vitamin D food supplements are allowed.
* Current evidence of clinically significant corneal (including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and keratoconjunctivitis) or retinal disorder (including but not limited to macular/retinal degeneration, diabetic retinopathy, and retinal detachment) as confirmed by ophthalmologic examination.
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to investigational product (IP) or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.7.4. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at Cycle 7 per IWG Response Criteria in subjects with R/R MCL. | 8 months
  To assess the efficacy of pemigatinib in subjects with R/R MCL.
To determine the ORR at Cycle 7 per IWG Response Criteria in subjects with R/R MZL. | 8 months
  To assess the efficacy of pemigatinib in subjects with R/R MZL.

SECONDARY OUTCOMES:
Complete Response (CR) rate at Cycle 7 per IWG Response Criteria. | 8 months
  To assess the CR rate at Cycle 7.
Duration of response (DoR), defined as the interval of time from the date of initial documented response (PR or better per IWG Response Criteria) to the time of progression from the best response, the start of a new therapy, or death from any cause. | 4 years
  To assess the DoR of the study population.
Progression-free survival (PFS) as defined as the time from study drug initiation to the time documented disease progression (as assessed by IWG Response Criteria), or death from any cause. | 4 years
  To assess median and 2 year PFS.
Overall survival (OS) as defined as the time from registration until death from any cause. | 4 years
  To assess median and 2 year OS in this study population.

CONTACTS AND LOCATIONS:
Overall Officials: Narendranath Epperla, MD, MS, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No